CLINICAL TRIAL: NCT01685437
Title: A Phase 3, Open-label Study of the Safety and Effectiveness of AA4500 Administered Twice Per Treatment Cycle for up to Four Treatment Cycles (2 x 4) in Men With Peyronie's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AUX-CC-806
Record Dates: First submitted 2012-09-12; First posted 2012-09-14 (Estimated); Results first posted 2015-04-07 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Peyronie's Disease
Keywords: Peyronie's disease, penile plaque, penile curvature
MeSH Terms: conditions — Penile Induration | interventions — Microbial Collagenase; xiapex

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AA4500 (Experimental): collagenase clostridium histolyticum
  Interventions: Biological: AA4500

INTERVENTIONS:
Biological: AA4500 — 2 injections separated by approximately 24 hours to 72 hours, repeated after 42 days (± 5 days) for up to 4 treatment cycles
  Other Names: Xiaflex; Xiapex

SUMMARY:
This study is a Phase 3, open-label study of the safety and efficacy of AA4500 0.58 mg in subjects with Peyronie's disease. Subjects will be screened for study eligibility within 21 days before the initial injection of study drug in the first treatment cycle. Enrollment will include all subjects who meet the eligibility criteria and who received placebo and completed one of the Auxilium-sponsored studies AUX-CC-803 or AUX-CC-804.

DETAILED DESCRIPTION:
After the final injection of each treatment cycle, the investigator or qualified designee (ie, qualified by license, education, and training to perform the study procedure according to local, state, and country requirements) will model the plaque in an attempt to stretch or elongate the plaque. If the subject's penile curvature is reduced to <15° after the first, second, or third cycle of injections or if the investigator determines further treatment is not clinically indicated (eg, adverse events; allergic reaction), subsequent treatment cycles will not be administered. Following the maximum of four treatment cycles, each subject will be followed for additional safety and efficacy assessments on Days 168 (± 7 days) and 252 (± 7 days) (nominal weeks 24 and 36).

ELIGIBILITY:
Inclusion Criteria:

No subject should be enrolled until all eligibility criteria have been satisfied. Subjects who completed their participation in Auxilium-sponsored studies AUX-CC-803 or AUX-CC-804 and received placebo in that study may enroll in this study provided they continue to meet the eligibility requirements. To qualify for the study a subject must:

1. Have penile curvature of at least 30° in the dorsal, lateral, or dorsal/lateral plane at screening. It must be possible to delineate the single plane of maximal curvature for evaluation during the study
2. Be judged to be in good health, based upon the results of a medical history, physical examination,and laboratory profile
3. Have participated in Study AUX-CC-803 or Study AUX-CC-804, received placebo in that study,and completed that study
4. Voluntarily sign and date an informed consent agreement approved by the Institutional Review Board/Independent Ethics Committee (IRB/IEC). The subject must also sign an authorization form to allow disclosure of his protected health information (PHI). The PHI authorization form and informed consent form may be an integrated form or may be separate forms depending on the institution
5. Be able to read, complete and understand the various rating instruments in English.

Exclusion Criteria:

A subject will be excluded from study participation if he:

1. Has a penile curvature of less than 30° or greater than 90° at the screening visit
2. Has any of the following conditions:

   * Chordee in the presence or absence of hypospadias
   * Thrombosis of the dorsal penile artery and/or vein
   * Infiltration by a benign or malignant mass resulting in penile curvature
   * Infiltration by an infectious agent, such as lymphogranuloma venereum
   * Ventral curvature from any cause
   * Presence of an active sexually transmitted disease
   * Known active hepatitis B or C
   * Known immune deficiency disease or be positive for human immunodeficiency virus (HIV)
3. Has previously undergone surgery for Peyronie's disease
4. Fails to have an erection which in the opinion of the investigator is sufficient to accurately measure the subject's penile deformity after administration of prostaglandin E1 or trimix or another suitable injectable pharmacologic stimulant according to the standard practice at the investigator's institution
5. Has a calcified plaque as evident by appropriate radiographic evaluation, penile x-ray or penile ultrasound that would prevent proper injection of study medication. Non-contiguous stippling of calcium is acceptable for inclusion provided the calcium deposit does not interfere with the injection of AA4500 into the plaque
6. Has an isolated hourglass deformity of the penis
7. Has the plaque causing curvature of the penis located proximal to the base of the penis, so that the injection of the local anesthetic would interfere with the injection of AA4500 into the plaque
8. Has previously received alternative medical therapies for Peyronie's disease administered by the intralesional route (including, but not limited to, steroids, verapamil, and the naturally occurring low molecular weight protein, interferon-α2b) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
9. Has received alternative medical therapies for Peyronie's disease administered by the oral (including, but not limited to, vitamin E [>500 U], potassium aminobenzoate [Potaba], tamoxifen, colchicine, and pentoxifylline, ,) or topical routes (including, but not limited to, verapamil applied as a cream) within 3 months before the first dose of study drug or plans to use any of these medical therapies at any time during the study
10. Has had extracorporeal shock wave therapy (ESWT) for the correction of Peyronie's disease within the 6-month period before screening or plans to have ESWT at any time during the study
11. Has used any mechanical type device for correction of Peyronie's disease within the 2-week period before screening or plans to use any these devices at any time during the study
12. Has used a mechanical device to induce a passive erection within the 2-week period before screening or plans to use any of these devices at any time during the study
13. Has significant erectile dysfunction that has failed to respond to oral treatment with phosphodiesterase type 5 (PDE5) inhibitors
14. Has a penile Duplex Doppler ultrasound evaluation at screening that shows compromised penile hemodynamics that in the opinion of the investigator is clinically significant
15. Has uncontrolled hypertension, as determined by the investigator
16. Has a known recent history of stroke, bleeding, or other significant medical condition, which in the investigator's opinion would make the subject unsuitable for enrollment in the study
17. Has received an investigational drug or treatment within 30 days before the first dose of study drug, except for placebo in Studies AUX-CC-803 or AUX-CC-804
18. Has a known systemic allergy to collagenase or any other excipient of AA4500
19. Has a known allergy to any concomitant medication required as per the protocol
20. Has received anticoagulant medication (except for ≤ 150 mg aspirin daily) during the 7 days before each dose of study drug
21. Has received any collagenase treatments within 30 days of the first dose of study drug
22. Has, at any time, received AA4500 for the treatment of Peyronie's disease
23. Is unwilling or unable to cooperate with the requirements of the study including completion of all scheduled study visits

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 189 (Actual)
Dates: Start 2012-09; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Kaufman, MD, Study Director — Auxilium Pharmaceuticals, Inc.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | AA4500
Started | 189
Completed | 158
Not Completed | 31
Not completed — Withdrawal by Subject | 22
Not completed — Lost to Follow-up | 3
Not completed — Adverse Event | 1
Not completed — Protocol Violation | 4
Not completed — Unable to make visits due to work | 1

BASELINE CHARACTERISTICS:
Arm/Group | AA4500
Number analyzed (Participants) | 189
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 134
  >=65 years | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.2 (7.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 189
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 184
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 1
  White | 186
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 162
  Australia | 27

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change From Baseline in Penile Curvature
Description: A negative value in the percentage change from baseline in penile curvature deformity (angle measured in degrees) indicates less curvature.
Time Frame: Baseline and Week 36
Population: Efficacy is based on modified intent-to-treat (mITT) population.
Measure: Mean (Standard Deviation); unit: percentage of curvature change
Arm/Group | AA4500
Number analyzed (Participants) | 126
percentage of curvature change | -36.3 (30.72)

2. Primary Outcome: Change From Baseline in the Peyronie's Disease Bother Domain of the Peyronie's Disease Questionnaire (PDQ)
Description: Peyronie's disease bother score range 0 (no issue or not at all bothered) to 4 (extremely bothered) on 4 questions; total score range 0 to 16. A decrease in the change from baseline total score in the Peyronie's disease bother domain of the PDQ is indicated by a negative number.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 126
units on a scale | -2.4 (3.34)

3. Secondary Outcome: Change From Baseline in the Severity of Peyronie's Disease Symptoms Domain of the PDQ
Description: Peyronie's disease symptoms (physical and psychological) severity score range 0 (none) to 4 (very severe) on 6 questions; total score range 0 to 24. A decrease in the change from baseline total score in the Peyronie's disease symptoms domain of the PDQ is indicated by a negative number.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 126
units on a scale | -2.9 (4.76)

4. Secondary Outcome: Change From Baseline in the Penile Pain Domain of the PDQ in Subjects With Baseline Penile Pain Score ≥4
Description: Penile pain scale range 0 (no pain) to 10 (extreme pain) on 3 questions; total score range 0 to 30. A decrease in the change from baseline total score in the penile pain domain of the PDQ is indicated by a negative number. Subjects were required to have a penile pain score of 4 or greater at baseline.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population; this population only includes those subjects in the mITT population with a baseline penile pain score of 4 or greater.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 36
units on a scale | -4.5 (4.75)

5. Secondary Outcome: A Responder Analysis Based on Subject Overall Global Assessment
Description: Subject overall global assessment of Peyronie's disease score range -3 (much worse) to 3 (much improved). A score of 1 (improved in a small but important way), 2 (moderately improved), or 3 indicate a responder.
Time Frame: Week 36
Population: Efficacy is based on the mITT population.
Measure: Number; unit: participants
Arm/Group | AA4500
Number analyzed (Participants) | 126
participants
  Responder Status - No | 32
  Responder Status - Yes | 94

6. Secondary Outcome: Change in the Overall Satisfaction Domain of the International Index of Erectile Function (IIEF)
Description: Overall satisfaction domain of the IIEF score range 0 to 5 on 2 questions where higher scores indicate improved function or satisfaction; total score range 0 to 10.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 126
units on a scale | 0.7 (2.13)

7. Secondary Outcome: Change From Baseline in Penile Plaque Consistency
Description: Penile plaque consistency score range 1 (non-palpable) to 5 (hard). A decrease in the change from baseline in penile plaque consistency is indicated by a negative number.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AA4500
Number analyzed (Participants) | 126
units on a scale | -0.4 (0.81)

8. Secondary Outcome: A Composite Responder Analysis Based on Change From Baseline in Penile Curvature and in the Peyronie's Disease Bother Score
Description: A composite responder is indicated by
  * a percent reduction from baseline in penile curvature greater than or equal to the threshold, and
  * a reduction from baseline in Peyronie's disease bother score greater than or equal to the threshold, or change in the overall sexual activity within the last 3 months to having vaginal intercourse from no vaginal intercourse at screening.
Time Frame: Week 36
Population: Composite responder analysis is based on the intent-to-treat (ITT) population.
Measure: Number; unit: participants
Arm/Group | AA4500
Number analyzed (Participants) | 189
participants
  No | 85
  Yes | 83
  Missing | 21

9. Secondary Outcome: Change From Baseline in Penile Length
Description: A negative value represents a reduction in measurement from baseline.
Time Frame: Baseline and Week 36
Population: Efficacy is based on the mITT population.
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | AA4500
Number analyzed (Participants) | 126
centimeters | 0.2 (1.16)

ADVERSE EVENTS:
Arm/Group | AA4500
Serious Adverse Events (participants affected / at risk) | 3/189
Other Adverse Events (participants affected / at risk) | 178/189
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=189)
Acoustic neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Caecitis (Gastrointestinal disorders) | 1 (1)
Calculus ureteric (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AA4500 (N=189)
Penile haematoma (Reproductive system and breast disorders) | 114 (271)
Penile pain (Reproductive system and breast disorders) | 64 (121)
Penile swelling (Reproductive system and breast disorders) | 57 (99)
Penile oedema (Reproductive system and breast disorders) | 46 (91)
Penile haemorrhage (Reproductive system and breast disorders) | 39 (73)
Injection site haematoma (General disorders) | 35 (66)
Injection site pain (General disorders) | 32 (50)
Injection site haemorrhage (General disorders) | 21 (56)
Injection site swelling (General disorders) | 20 (27)
Contusion (Injury, poisoning and procedural complications) | 17 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other